CLINICAL TRIAL: NCT04880746
Title: Efficacy and Safety of Cladribine Combined With BEAC ( Semustine, Etoposide, Cytarabine, Cyclophosphamide) Pretreatment Regimen in the Treatment of Peripheral T-cell Lymphoma: a Multicenter Clinical Study
Brief Title: Efficacy and Safety of Cladribine Combined With BEAC Pretreatment Regimen in the Treatment of Peripheral T-cell Lymphoma: a Multicenter Clinical Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Xinqiao Hospital of Chongqing (Other); The First Affiliated Hospital of Anhui Medical University (Other); Harbin Hematology and Oncology Institute (Other); Affiliated Zhongshan Hospital of Dalian University (Other); Qilu Hospital of Shandong University (Other); Fujian Medical University Union Hospital (Other); Shanxi Province Cancer Hospital (Other); RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director, Hematology Department, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCT-001
Record Dates: First submitted 2021-04-17; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell lymphoma; Autologous stem cell transplantation; Cladribine; BEAC
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — BAEC protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEAC (Active Comparator): Patients in this arm will receive BEAC (Semustine, Etoposide, Cytarabine, Cyclophosphamide) as pretreatment regimen of ASCT
  Interventions: Drug: BEAC
- Cladribine combined with BEAC (Experimental): Patients in this arm will receive Cladribine combined with BEAC (Semustine, Etoposide, Cytarabine, Cyclophosphamide) as pretreatment regimen of ASCT
  Interventions: Drug: Cladribine combined with BEAC

INTERVENTIONS:
Drug: BEAC — Semustine, 300 mg/m2，-6d； Etoposide, 100 mg/m2，-5～-2d； Cytarabine, 100mg/m2，q12h，-5～-2d； Cyclophosphamide, 1.5g/m2，-5～-2d
  Arms: BEAC
Drug: Cladribine combined with BEAC — Cladribine, 6mg/m2，-5～-2d, two hours before Cytarabine Semustine, 300 mg/m2，-6d； Etoposide, 100 mg/m2，-5～-2d； Cytarabine, 100mg/m2，q12h，-5～-2d； Cyclophosphamide, 1.5g/m2，-5～-2d
  Arms: Cladribine combined with BEAC

SUMMARY:
This multi-center clinical study will evaluate the efficacy and safety of Cladribine Combined With BEAC Pretreatment Regimen in the Treatment of Peripheral T-cell Lymphoma.

DETAILED DESCRIPTION:
Peripheral T-cell lymphomas (PTCL) is a group of highly heterogeneous aggressive non-Hodgkin lymphomas originating from mature post-thymic T lymphocytes or NK/T cells. The treatment effect of patients receiving autologous hematopoietic stem cell transplantation (ASCT) is better than traditional chemotherapy, but the recurrence after transplantation is still as high as 50%. It is an urgent clinical problem to reduce the recurrence after PTCL transplantation. Cladribine can kill quiescent tumor cells, which is the main reason of tumor recurrence. Since 2018, our center has used cladribine combined with BEAC pretreatment regimen to treat 20 patients with PTCL. The PFS reached 68% at 2 years, which is about 15% higher than the previous classic BEAC regimen. This multi-center clinical study will further evaluate the efficacy and safety of Cladribine combined with BEAC pretreatment regimen in the Treatment of Peripheral T-cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old, no gender limit;
* ECOG 0-2, estimated survival time ≥ 3 months;
* Pathologically newly diagnosed with PTCL (except ALK+ anaplastic large cell lymphoma), with PR or CR after 6 cycles of induction chemotherapy;
* Hb≥80g/L, ANC≥1.0×10^9/L, PLT≥75×10^9/L; TBIL≤1.5×ULN, ALT/AST≤2.0× ULN, Cr ≤1.5×ULN in the 14 days before enrollment
* Have not received hematopoietic stem cell transplantation and other treatments within 4 weeks before enrollment;
* The number of hematopoietic stem cells requires MNC ≥3×10^8/kg and/or CD34 cells ≥2×10^6/kg;
* Informed consented

Exclusion Criteria:

* Accompanied by severe cardiac insufficiency, cardiac ejection fraction <60%; or severe arrhythmia, intolerance of pretreatment;
* Accompanied by severe pulmonary insufficiency (obstructive and or restrictive ventilatory disorders), intolerance of pretreatment;
* Accompanied by severe liver function impairment, liver function indexes (ALT, TBIL) are more than 3 times higher than the upper limit of normal, intolerance of pretreatment;
* Accompanied by severe renal insufficiency, the renal function index (Cr) is more than 2 times the upper limit of normal; or the 24-hour urine creatinine clearance rate Ccr is less than 50ml/min, intolerance of pretreatment;
* Severe active infection before transplantation, intolerance of pretreatment;
* Accompanied by brain dysfunction or severe mental illness, unable to understand or follow the research plan;
* Pregnant or lactation；
* Accompanied by other malignant tumors in need of treatment;
* Patients who cannot guarantee the completion of the necessary treatment plan and follow-up observation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2020-10-17 (Actual); Primary Completion 2024-10-17 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of ASCT until the date of the first documented day of disease progression or relapse, using Revised Standards for Efficacy Evaluation of Malignant Lymphoma in 2007, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | Baseline up to data cut-off (up to approximately 2 years)
  Overall survival was defined as the time from the date of ASCT to the date of death from any cause.
Overall remission rate | 3 months after the transplantation
  Percentage of participants with overall response was determined on the basis of Revised Standards for Efficacy Evaluation of Malignant Lymphoma in 2007.
Transplantation-related adverse reactions | Baseline up to data cut-off (up to approximately 5 years)
  Transplantation-related adverse reactions are any untoward medical occurrence in a participant which is related to ASCT
Patient tolerance | Through the whole course of ASCT, an average of one month
  Percentage of participants who can tolerate the whole treatment of ASCT
Relapse rate | Baseline up to data cut-off (up to approximately 5 years)
  Percentage of participants who relapse determined on the basis of Revised Standards for Efficacy Evaluation of Malignant Lymphoma in 2007.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No